CLINICAL TRIAL: NCT07078136
Title: Multicenter Observational Study of a Multimodal AI Model Using EUS, White-Light Endoscopy, and Clinical Data for Diagnosis of Upper GI Mesenchymal Tumors and Risk Stratification of Gastric GISTs
Brief Title: Multicenter Observational Study of Multimodal AI for Upper GI Mesenchymal Tumor Diagnosis
Status: Recruiting | Type: Observational
Sponsor: Huazhong University of Science and Technology (Other)
Responsible Party: Principal Investigator, Bin Cheng, Professor, Huazhong University of Science and Technology
Other Study IDs: GIST-AI 2025
Record Dates: First submitted 2025-07-02; First posted 2025-07-22 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Submucosal Tumor; Gastrointestinal Stromal Tumor (GIST); Leiomyoma; Schwannoma
Keywords: Artificial Intelligence; Endoscopic ultrasound; white-light endoscopy
MeSH Terms: conditions — Gastrointestinal Stromal Tumors; Leiomyoma; Neurilemmoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All Participants: All enrolled patients with upper gastrointestinal subepithelial lesions confirmed by histopathology. Each participant will undergo standard diagnostic evaluation and independent multimodal AI prediction and expert endoscopist diagnosis.
  Interventions: Diagnostic Test: Multimodal AI Model; Diagnostic Test: Expert Endoscopist Assessment

INTERVENTIONS:
Diagnostic Test: Multimodal AI Model — Patients' endoscopic images, EUS images, and clinical data will be analyzed by a multimodal AI model for lesion classification and GIST risk stratification.
Diagnostic Test: Expert Endoscopist Assessment — Endoscopic ultrasound images will be interpreted by experienced endoscopists for comparison with the AI model.

SUMMARY:
This study develops a multimodal AI model using endoscopic ultrasound, white-light endoscopy, and clinical information to support the diagnosis of upper GI mesenchymal tumors and the risk stratification of gastric GISTs.

DETAILED DESCRIPTION:
This is a multicenter, observational study designed to evaluate the diagnostic performance of a multimodal artificial intelligence (AI) model for the classification of upper gastrointestinal subepithelial lesions (SELs) and risk stratification of gastric gastrointestinal stromal tumors (gGISTs). The study combines retrospective image data for training and validation with prospectively recruited cases for testing.

Endoscopic ultrasound (EUS) images, white-light endoscopy (WLE) images, and relevant clinical data will be collected according to strict image quality control criteria. The multimodal AI model integrates these inputs using a multi-branch fusion strategy. A cross-validation trial will be conducted using prospectively recruited patients' data from multiple centers to compare the diagnostic and predictive performance of endoscopists with and without AI assistance for both lesion classification and risk stratification.

According to existing literature, no multimodal AI model has yet reported diagnostic performance for classifying SELs or for risk stratification of gastric gGISTs. It is assumed that the multimodal AI model will achieve a diagnostic accuracy of 95% for classifying upper gastrointestinal SELs and 95% for gGIST risk stratification. In comparison, the diagnostic accuracy of endoscopists is approximately 73.3%-75% for differentiating GIST from non-GIST and 72.4%-78.9% for risk stratification of gGISTs . GISTs account for about 67-68% of all lesions . Using a two-sided confidence interval with α = 0.05 and β = 0.2, and considering a 20% potential dropout rate, the minimum sample size required for prospective SEL classification is 65 cases, and 88 gGIST cases for risk stratification. Since the risk stratification task requires a larger sample size and GISTs are the common target of both tasks, the final planned sample size is 130 patients with upper GI SELs, which meets the statistical requirements for all primary endpoints.

The study team will screen patients based on the inclusion and exclusion criteria, ensure that all required examinations are completed to confirm eligibility, and record pre-treatment test results. All prospective participants will provide written informed consent before any study-related examinations.

This study is purely observational. No additional interventions will be performed on participants, nor will any additional costs be incurred. Patients' access to optimal diagnostic or treatment options will not be affected. The primary potential risk is the breach of patient privacy; the research team will establish a strict data security and monitoring plan and inform participants that their data will be used for clinical research purposes.

This study is purely observational. No additional interventions will be performed on participants, nor will any additional costs be incurred. Patients' access to optimal diagnostic or treatment options will not be affected. The primary potential risk is the breach of patient privacy; the research team will establish a strict data security and monitoring plan and inform participants that their data will be used for clinical research purposes.

Each enrolled participant will undergo diagnostic assessment by both the multimodal AI model and expert endoscopists. The AI model and expert interpretation will be blinded to each other. Final diagnosis will be confirmed by histopathology. Diagnostic performance will be compared using paired analysis. All statistical tests will be two-sided, and differences will be considered statistically significant at P < 0.05. Continuous variables will be described as mean ± standard deviation. Categorical variables will be presented as counts and percentages. (1) Diagnostic Performance: The diagnostic performance of endoscopists and the AI model will be compared using sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), accuracy, and area under the curve (AUC). F1-score (harmonic mean) and balanced accuracy will be calculated to address class imbalance (e.g., GIST vs. other lesions). (2) Continuous Data: Comparisons with baseline values will be conducted using paired t-tests, ANOVA, or rank-sum tests as appropriate. (3) Categorical Data: Group comparisons will use Chi-square tests (including CMH Chi-square test) or Fisher's exact test. (4) Baseline Comparability: Demographic and baseline characteristics will be compared using independent t-tests or Chi-square tests to assess group balance. (5) Effectiveness Analysis: The primary effectiveness endpoint is the diagnostic accuracy for GI subepithelial lesions. The difference in proportions and Youden index will be compared using the approximate normal Z test or Chi-square test with center effect control. (6) Software: All statistical analyses will be performed using SPSS version 26.0.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years old
* Patients with an upper gastrointestinal subepithelial lesion (SEL) identified by white-light endoscopy and who have completed an endoscopic ultrasound (EUS) examination
* Patients with a histopathological diagnosis of GIST confirmed by surgical or endoscopic resection, or other SELs confirmed by surgical resection, EUS-guided sampling, or other biopsy techniques
* EUS image quality meets the following quality control standards

  1. Equipment requirements: Olympus EU-ME2/ME1 processor (Olympus Medical Systems Corp., Tokyo, Japan); radial EUS scope (GF-UE260/GF-UE240; Olympus, Tokyo, Japan) or linear EUS scope (GF-UCT260/GF-UCT240; Olympus, Tokyo, Japan); miniature probe (UM2R/3R; Olympus, Tokyo, Japan); Pentax ARIETTA 850 processor (Pentax, Tokyo, Japan); radial EUS scope (EG-3670URK, Pentax, Tokyo, Japan); linear EUS scope (EG-3870UT, Pentax, Tokyo, Japan); Fujifilm SU-8000 or SU-9000 processor; linear EUS scope (EG-580UT, Fujifilm, Tokyo, Japan); radial EUS scope (EG-580UR, Fujifilm, Tokyo, Japan)
  2. EUS images clearly showing the lesion and surrounding tissue characteristics (at least 5 images or video); must include at least one image of the maximum lesion diameter, one image showing the layer of origin, and one image demonstrating the growth pattern (intraluminal/extraluminal)
  3. EUS images must not contain artificial annotations, such as measurement scales, biopsy needles, Doppler signals, or elastography overlays
  4. Image resolution must be at least 448 × 448 pixels
* WLE (white-light endoscopy) image quality meets the following standards: images must clearly show the lesion location, mucosal features, and margins; at least one close-up and one distant view
* Complete clinical data and histopathological reports must be available

Exclusion Criteria:

* Age < 18 years old
* Absolute contraindications for EUS examination, history of gastric surgery, pregnancy, severe comorbidities, or known allergy to anesthetic agents
* EUS examination terminated prematurely due to esophageal stricture, obstruction, large space-occupying lesions, rapid changes in heart rate or respiratory rate, patient intolerance, or excessive residual food
* EUS image quality does not meet the required quality control standards
* Pathological specimens do not meet diagnostic requirements: insufficient biopsy tissue (only R0 resection specimens are accepted for the GIST group), or incomplete immunohistochemical staining (missing CD117/CD34/DOG-1 expression report for the GIST group)
* Pathological results indicate that the lesion is a metastatic tumor originating from another site

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The cohort will be selected from several hospitals in China, including Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology.
Sampling Method: Non-Probability Sample
Enrollment: 130 (Estimated)
Dates: Start 2025-07-28 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Diagnostic accuracy of a multimodal AI model for differentiating gastrointestinal stromal tumors (GISTs) from other upper gastrointestinal mesenchymal tumors | After the training process of the multimodal AI model is completed，on average per year
  Receiver operating characteristic (ROC) analyses, sensitivity, specificity, accuracy, positive predictive value and negative predictive value will be used to evaluate the efficacy of the model
Predictive accuracy of the multimodal AI model for risk stratification of GISTs | After the training process of the multimodal AI model is completed，on average per year
  ROC analyses, sensitivity, specificity, accuracy, positive predictive value and negative predictive value will be used to evaluate the efficacy of the model

SECONDARY OUTCOMES:
Comparison of Diagnostic Accuracy Between the Multimodal AI Model and Single-Modality Models | After the training process of the Multimodal AI model is completed，on average per year
  Receiver operating characteristic (ROC) analyses, sensitivity, specificity, accuracy, positive predictive value and negative predictive value will be used to evaluate the efficacy of the model
Comparison of diagnostic accuracy between the multimodal AI model and experienced endoscopists for differentiating GISTs and non-GIST mesenchymal tumors | After the testing process of the multimodal AI model is completed，on average per year
  The diagnostic accuracy of the AI model and expert endoscopists will be compared within the same participants, using histopathology as the gold standard. Receiver operating characteristic (ROC) analyses, sensitivity, specificity, accuracy, positive predictive value and negative predictive value will be used to evaluate the efficacy of the model
Comparison of the predictive accuracy for GIST risk stratification between the multimodal AI model and experienced endoscopists | After the testing process of the multimodal AI model is completed，on average per year
  The diagnostic accuracy of the AI model and expert endoscopists will be compared within the same participants, using histopathology as the gold standard. Receiver operating characteristic (ROC) analyses, sensitivity, specificity, accuracy, positive predictive value and negative predictive value will be used to evaluate the efficacy of the model

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chinese Society of Digestive Endoscopy Tunnel Technology Collaboration Group, Endoscopist Branch of Chinese Medical Doctor Association, and Digestive Endoscopy Branch of Beijing Medical Association. Expert Consensus on Endoscopic Diagnosis and Treatment of Gastrointestinal Stromal Tumors in China (2020, Beijing). Chinese Journal of Digestive Endoscopy, 2021(07): 505-514.
- [Background] Shen L, Cao H, Qin S, et al. Chinese Consensus on the Diagnosis and Treatment of Gastrointestinal Stromal Tumors (2017 Version). Electronic Journal of Integrated Cancer Therapy, 2018; 4(01): 31-43.
- [Background] Gomes RSA, de Oliveira GHP, de Moura DTH, Kotinda APST, Matsubayashi CO, Hirsch BS, Veras MO, Ribeiro Jordao Sasso JG, Trasolini RP, Bernardo WM, de Moura EGH. Endoscopic ultrasound artificial intelligence-assisted for prediction of gastrointestinal stromal tumors diagnosis: A systematic review and meta-analysis. World J Gastrointest Endosc. 2023 Aug 16;15(8):528-539. doi: 10.4253/wjge.v15.i8.528. PMID 37663113
- [Result] Abe K, Tominaga K, Yamamiya A, Inaba Y, Kanamori A, Kondo M, Suzuki T, Watanabe H, Kawano M, Sato T, Yoshitake N, Ohwada T, Konno M, Hanatsuka K, Masuyama H, Goda K, Haruyama Y, Irisawa A; NUTSHELL20 Study group. Natural History of Small Gastric Subepithelial Lesions Less than 20 mm: A Multicenter Retrospective Observational Study (NUTSHELL20 Study). Digestion. 2023;104(3):174-186. doi: 10.1159/000527421. Epub 2022 Dec 5. PMID 36470211
- [Result] Standards of Practice Committee; Faulx AL, Kothari S, Acosta RD, Agrawal D, Bruining DH, Chandrasekhara V, Eloubeidi MA, Fanelli RD, Gurudu SR, Khashab MA, Lightdale JR, Muthusamy VR, Shaukat A, Qumseya BJ, Wang A, Wani SB, Yang J, DeWitt JM. The role of endoscopy in subepithelial lesions of the GI tract. Gastrointest Endosc. 2017 Jun;85(6):1117-1132. doi: 10.1016/j.gie.2017.02.022. Epub 2017 Apr 3. No abstract available. PMID 28385194
- [Result] Li J, Ye Y, Wang J, Zhang B, Qin S, Shi Y, He Y, Liang X, Liu X, Zhou Y, Wu X, Zhang X, Wang M, Gao Z, Lin T, Cao H, Shen L, Chinese Society Of Clinical Oncology Csco Expert Committee On Gastrointestinal Stromal Tumor. Chinese consensus guidelines for diagnosis and management of gastrointestinal stromal tumor. Chin J Cancer Res. 2017 Aug;29(4):281-293. doi: 10.21147/j.issn.1000-9604.2017.04.01. PMID 28947860
- [Result] Miettinen M, Sobin LH, Lasota J. Gastrointestinal stromal tumors of the stomach: a clinicopathologic, immunohistochemical, and molecular genetic study of 1765 cases with long-term follow-up. Am J Surg Pathol. 2005 Jan;29(1):52-68. doi: 10.1097/01.pas.0000146010.92933.de. PMID 15613856
- [Result] Kawanowa K, Sakuma Y, Sakurai S, Hishima T, Iwasaki Y, Saito K, Hosoya Y, Nakajima T, Funata N. High incidence of microscopic gastrointestinal stromal tumors in the stomach. Hum Pathol. 2006 Dec;37(12):1527-35. doi: 10.1016/j.humpath.2006.07.002. Epub 2006 Sep 25. PMID 16996566
- [Result] Pang T, Zhao Y, Fan T, Hu Q, Raymond D, Cao S, Zhang W, Wang Y, Zhang B, Lv Y, Zhang X, Ling T, Zhuge Y, Wang L, Zou X, Huang Q, Xu G. Comparison of Safety and Outcomes between Endoscopic and Surgical Resections of Small (</= 5 cm) Primary Gastric Gastrointestinal Stromal Tumors. J Cancer. 2019 Jul 10;10(17):4132-4141. doi: 10.7150/jca.29443. eCollection 2019. PMID 31417658
- [Result] Coe TM, Fero KE, Fanta PT, Mallory RJ, Tang CM, Murphy JD, Sicklick JK. Population-Based Epidemiology and Mortality of Small Malignant Gastrointestinal Stromal Tumors in the USA. J Gastrointest Surg. 2016 Jun;20(6):1132-40. doi: 10.1007/s11605-016-3134-y. Epub 2016 Mar 29. PMID 27025710
- [Result] Nishida T, Blay JY, Hirota S, Kitagawa Y, Kang YK. The standard diagnosis, treatment, and follow-up of gastrointestinal stromal tumors based on guidelines. Gastric Cancer. 2016 Jan;19(1):3-14. doi: 10.1007/s10120-015-0526-8. Epub 2015 Aug 15. PMID 26276366
- [Result] Casali PG, Abecassis N, Aro HT, Bauer S, Biagini R, Bielack S, Bonvalot S, Boukovinas I, Bovee JVMG, Brodowicz T, Broto JM, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dileo P, Eriksson M, Fedenko A, Ferraresi V, Ferrari A, Ferrari S, Frezza AM, Gasperoni S, Gelderblom H, Gil T, Grignani G, Gronchi A, Haas RL, Hassan B, Hohenberger P, Issels R, Joensuu H, Jones RL, Judson I, Jutte P, Kaal S, Kasper B, Kopeckova K, Krakorova DA, Le Cesne A, Lugowska I, Merimsky O, Montemurro M, Pantaleo MA, Piana R, Picci P, Piperno-Neumann S, Pousa AL, Reichardt P, Robinson MH, Rutkowski P, Safwat AA, Schoffski P, Sleijfer S, Stacchiotti S, Sundby Hall K, Unk M, Van Coevorden F, van der Graaf WTA, Whelan J, Wardelmann E, Zaikova O, Blay JY; ESMO Guidelines Committee and EURACAN. Gastrointestinal stromal tumours: ESMO-EURACAN Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2018 Oct 1;29(Suppl 4):iv267. doi: 10.1093/annonc/mdy320. No abstract available. PMID 30188977
- [Result] von Mehren M, Randall RL, Benjamin RS, Boles S, Bui MM, Conrad EU 3rd, Ganjoo KN, George S, Gonzalez RJ, Heslin MJ, Kane JM 3rd, Koon H, Mayerson J, McCarter M, McGarry SV, Meyer C, O'Donnell RJ, Pappo AS, Paz IB, Petersen IA, Pfeifer JD, Riedel RF, Schuetze S, Schupak KD, Schwartz HS, Tap WD, Wayne JD, Bergman MA, Scavone J. Soft Tissue Sarcoma, Version 2.2016, NCCN Clinical Practice Guidelines in Oncology. J Natl Compr Canc Netw. 2016 Jun;14(6):758-86. doi: 10.6004/jnccn.2016.0078. PMID 27283169
- [Result] Nishida T, Hirota S, Yanagisawa A, Sugino Y, Minami M, Yamamura Y, Otani Y, Shimada Y, Takahashi F, Kubota T; GIST Guideline Subcommittee. Clinical practice guidelines for gastrointestinal stromal tumor (GIST) in Japan: English version. Int J Clin Oncol. 2008 Oct;13(5):416-30. doi: 10.1007/s10147-008-0798-7. Epub 2008 Oct 23. PMID 18946752
- [Result] Casali PG, Blay JY, Abecassis N, Bajpai J, Bauer S, Biagini R, Bielack S, Bonvalot S, Boukovinas I, Bovee JVMG, Boye K, Brodowicz T, Buonadonna A, De Alava E, Dei Tos AP, Del Muro XG, Dufresne A, Eriksson M, Fedenko A, Ferraresi V, Ferrari A, Frezza AM, Gasperoni S, Gelderblom H, Gouin F, Grignani G, Haas R, Hassan AB, Hindi N, Hohenberger P, Joensuu H, Jones RL, Jungels C, Jutte P, Kasper B, Kawai A, Kopeckova K, Krakorova DA, Le Cesne A, Le Grange F, Legius E, Leithner A, Lopez-Pousa A, Martin-Broto J, Merimsky O, Messiou C, Miah AB, Mir O, Montemurro M, Morosi C, Palmerini E, Pantaleo MA, Piana R, Piperno-Neumann S, Reichardt P, Rutkowski P, Safwat AA, Sangalli C, Sbaraglia M, Scheipl S, Schoffski P, Sleijfer S, Strauss D, Strauss SJ, Hall KS, Trama A, Unk M, van de Sande MAJ, van der Graaf WTA, van Houdt WJ, Frebourg T, Gronchi A, Stacchiotti S; ESMO Guidelines Committee, EURACAN and GENTURIS. Electronic address: clinicalguidelines@esmo.org. Gastrointestinal stromal tumours: ESMO-EURACAN-GENTURIS Clinical Practice Guidelines for diagnosis, treatment and follow-up. Ann Oncol. 2022 Jan;33(1):20-33. doi: 10.1016/j.annonc.2021.09.005. Epub 2021 Sep 21. No abstract available. PMID 34560242
- [Result] Baysal B, Masri OA, Eloubeidi MA, Senturk H. The role of EUS and EUS-guided FNA in the management of subepithelial lesions of the esophagus: A large, single-center experience. Endosc Ultrasound. 2017 Sep-Oct;6(5):308-316. doi: 10.4103/2303-9027.155772. PMID 26365993
- [Result] Daimaru Y, Kido H, Hashimoto H, Enjoji M. Benign schwannoma of the gastrointestinal tract: a clinicopathologic and immunohistochemical study. Hum Pathol. 1988 Mar;19(3):257-64. doi: 10.1016/s0046-8177(88)80518-5. PMID 3126126
- [Result] Mekras A, Krenn V, Perrakis A, Croner RS, Kalles V, Atamer C, Grutzmann R, Vassos N. Gastrointestinal schwannomas: a rare but important differential diagnosis of mesenchymal tumors of gastrointestinal tract. BMC Surg. 2018 Jul 25;18(1):47. doi: 10.1186/s12893-018-0379-2. PMID 30045739
- [Result] Lauricella S, Valeri S, Masciana G, Gallo IF, Mazzotta E, Pagnoni C, Costanza S, Falcone L, Benvenuto D, Caricato M, Capolupo GT. What About Gastric Schwannoma? A Review Article. J Gastrointest Cancer. 2021 Mar;52(1):57-67. doi: 10.1007/s12029-020-00456-2. PMID 32964322
- [Result] Karaca C, Turner BG, Cizginer S, Forcione D, Brugge W. Accuracy of EUS in the evaluation of small gastric subepithelial lesions. Gastrointest Endosc. 2010 Apr;71(4):722-7. doi: 10.1016/j.gie.2009.10.019. Epub 2010 Feb 19. PMID 20171632
- [Result] Hwang JH, Saunders MD, Rulyak SJ, Shaw S, Nietsch H, Kimmey MB. A prospective study comparing endoscopy and EUS in the evaluation of GI subepithelial masses. Gastrointest Endosc. 2005 Aug;62(2):202-8. doi: 10.1016/s0016-5107(05)01567-1. PMID 16046979
- [Result] Minoda Y, Chinen T, Osoegawa T, Itaba S, Haraguchi K, Akiho H, Aso A, Sumida Y, Komori K, Ogino H, Ihara E, Ogawa Y. Superiority of mucosal incision-assisted biopsy over ultrasound-guided fine needle aspiration biopsy in diagnosing small gastric subepithelial lesions: a propensity score matching analysis. BMC Gastroenterol. 2020 Jan 21;20(1):19. doi: 10.1186/s12876-020-1170-2. PMID 31964357
- [Result] de Moura DTH, McCarty TR, Jirapinyo P, Ribeiro IB, Flumignan VK, Najdawai F, Ryou M, Lee LS, Thompson CC. EUS-guided fine-needle biopsy sampling versus FNA in the diagnosis of subepithelial lesions: a large multicenter study. Gastrointest Endosc. 2020 Jul;92(1):108-119.e3. doi: 10.1016/j.gie.2020.02.021. Epub 2020 Feb 25. PMID 32105712
- [Result] Osoegawa T, Minoda Y, Ihara E, Komori K, Aso A, Goto A, Itaba S, Ogino H, Nakamura K, Harada N, Makihara K, Tsuruta S, Yamamoto H, Ogawa Y. Mucosal incision-assisted biopsy versus endoscopic ultrasound-guided fine-needle aspiration with a rapid on-site evaluation for gastric subepithelial lesions: A randomized cross-over study. Dig Endosc. 2019 Jul;31(4):413-421. doi: 10.1111/den.13367. Epub 2019 Apr 2. PMID 30723945
- [Result] Joensuu H. Risk stratification of patients diagnosed with gastrointestinal stromal tumor. Hum Pathol. 2008 Oct;39(10):1411-9. doi: 10.1016/j.humpath.2008.06.025. PMID 18774375
- [Result] Shah P, Gao F, Edmundowicz SA, Azar RR, Early DS. Predicting malignant potential of gastrointestinal stromal tumors using endoscopic ultrasound. Dig Dis Sci. 2009 Jun;54(6):1265-9. doi: 10.1007/s10620-008-0484-7. Epub 2008 Aug 29. PMID 18758957
- [Result] Chen T, Xu L, Dong X, Li Y, Yu J, Xiong W, Li G. The roles of CT and EUS in the preoperative evaluation of gastric gastrointestinal stromal tumors larger than 2 cm. Eur Radiol. 2019 May;29(5):2481-2489. doi: 10.1007/s00330-018-5945-6. Epub 2019 Jan 7. PMID 30617491
- [Result] Chen H, Xu Z, Huo J, Liu D. Submucosal tunneling endoscopic resection for simultaneous esophageal and cardia submucosal tumors originating from the muscularis propria layer (with video). Dig Endosc. 2015 Jan;27(1):155-8. doi: 10.1111/den.12227. Epub 2014 Jan 20. PMID 24444087
- [Result] He G, Wang J, Chen B, Xing X, Wang J, Chen J, He Y, Cui Y, Chen M. Feasibility of endoscopic submucosal dissection for upper gastrointestinal submucosal tumors treatment and value of endoscopic ultrasonography in pre-operation assess and post-operation follow-up: a prospective study of 224 cases in a single medical center. Surg Endosc. 2016 Oct;30(10):4206-13. doi: 10.1007/s00464-015-4729-1. Epub 2016 Jan 28. PMID 26823060
- [Result] Hirai K, Kuwahara T, Furukawa K, Kakushima N, Furune S, Yamamoto H, Marukawa T, Asai H, Matsui K, Sasaki Y, Sakai D, Yamada K, Nishikawa T, Hayashi D, Obayashi T, Komiyama T, Ishikawa E, Sawada T, Maeda K, Yamamura T, Ishikawa T, Ohno E, Nakamura M, Kawashima H, Ishigami M, Fujishiro M. Artificial intelligence-based diagnosis of upper gastrointestinal subepithelial lesions on endoscopic ultrasonography images. Gastric Cancer. 2022 Mar;25(2):382-391. doi: 10.1007/s10120-021-01261-x. Epub 2021 Nov 16. PMID 34783924
- [Result] Byrne MF, Chapados N, Soudan F, Oertel C, Linares Perez M, Kelly R, Iqbal N, Chandelier F, Rex DK. Real-time differentiation of adenomatous and hyperplastic diminutive colorectal polyps during analysis of unaltered videos of standard colonoscopy using a deep learning model. Gut. 2019 Jan;68(1):94-100. doi: 10.1136/gutjnl-2017-314547. Epub 2017 Oct 24. PMID 29066576
- [Result] Yang X, Wang H, Dong Q, Xu Y, Liu H, Ma X, Yan J, Li Q, Yang C, Li X. An artificial intelligence system for distinguishing between gastrointestinal stromal tumors and leiomyomas using endoscopic ultrasonography. Endoscopy. 2022 Mar;54(3):251-261. doi: 10.1055/a-1476-8931. Epub 2022 Jun 9. PMID 33827140
- [Result] Oh CK, Kim T, Cho YK, Cheung DY, Lee BI, Cho YS, Kim JI, Choi MG, Lee HH, Lee S. Convolutional neural network-based object detection model to identify gastrointestinal stromal tumors in endoscopic ultrasound images. J Gastroenterol Hepatol. 2021 Dec;36(12):3387-3394. doi: 10.1111/jgh.15653. Epub 2021 Aug 16. PMID 34369001
- [Result] Niikura R, Aoki T, Shichijo S, Yamada A, Kawahara T, Kato Y, Hirata Y, Hayakawa Y, Suzuki N, Ochi M, Hirasawa T, Tada T, Kawai T, Koike K. Artificial intelligence versus expert endoscopists for diagnosis of gastric cancer in patients who have undergone upper gastrointestinal endoscopy. Endoscopy. 2022 Aug;54(8):780-784. doi: 10.1055/a-1660-6500. Epub 2022 May 4. PMID 34607377
- [Result] Liu J, Huang J, Song Y, He Q, Fang W, Wang T, Zheng Z, Liu W. Differentiating Gastrointestinal Stromal Tumors From Leiomyomas of Upper Digestive Tract Using Convolutional Neural Network Model by Endoscopic Ultrasonography. J Clin Gastroenterol. 2024 Jul 1;58(6):574-579. doi: 10.1097/MCG.0000000000001907. PMID 37646533
- [Result] Lu Y, Chen L, Wu J, Er L, Shi H, Cheng W, Chen K, Liu Y, Qiu B, Xu Q, Feng Y, Tang N, Wan F, Sun J, Zhi M. Artificial intelligence in endoscopic ultrasonography: risk stratification of gastric gastrointestinal stromal tumors. Therap Adv Gastroenterol. 2023 May 30;16:17562848231177156. doi: 10.1177/17562848231177156. eCollection 2023. PMID 37274299
- [Result] Seven G, Silahtaroglu G, Kochan K, Ince AT, Arici DS, Senturk H. Use of Artificial Intelligence in the Prediction of Malignant Potential of Gastric Gastrointestinal Stromal Tumors. Dig Dis Sci. 2022 Jan;67(1):273-281. doi: 10.1007/s10620-021-06830-9. Epub 2021 Feb 6. PMID 33547537
- [Result] Kline A, Wang H, Li Y, Dennis S, Hutch M, Xu Z, Wang F, Cheng F, Luo Y. Multimodal machine learning in precision health: A scoping review. NPJ Digit Med. 2022 Nov 7;5(1):171. doi: 10.1038/s41746-022-00712-8. PMID 36344814
- [Result] Kim SY, Shim KN, Lee JH, Lim JY, Kim TO, Choe AR, Tae CH, Jung HK, Moon CM, Kim SE, Jung SA. Comparison of the Diagnostic Ability of Endoscopic Ultrasonography and Abdominopelvic Computed Tomography in the Diagnosis of Gastric Subepithelial Tumors. Clin Endosc. 2019 Nov;52(6):565-573. doi: 10.5946/ce.2019.019. Epub 2019 Jul 17. PMID 31311912
- [Result] Lefort C, Gupta V, Lisotti A, Palazzo L, Fusaroli P, Pujol B, Gincul R, Fumex F, Palazzo M, Napoleon B. Diagnosis of gastric submucosal tumors and estimation of malignant risk of GIST by endoscopic ultrasound. Comparison between B mode and contrast-harmonic mode. Dig Liver Dis. 2021 Nov;53(11):1486-1491. doi: 10.1016/j.dld.2021.06.013. Epub 2021 Jul 14. PMID 34272196